CLINICAL TRIAL: NCT05567029
Title: A Phase 1 Study in Healthy Subjects to Evaluate the Bioavailability of Risankizumab 150mg/mL Formulation in the 180 mg Prefilled Syringe Relative to 90mg/mL Formulation in the 90 mg Prefilled Syringe
Brief Title: Study to Evaluate the Relative Bioavailability of Two Risankizumab Drug Product Presentations in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M23-522
Record Dates: First submitted 2022-10-03; First posted 2022-10-05 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Healthy Volunteers
Keywords: Risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Risankizumab Dose A (Experimental): Participants will receive subcutaneous dose of risankizumab dose A.
  Interventions: Drug: Risankizumab Dose A
- Risankizumab Dose B (Experimental): Participants will receive subcutaneous dose of risankizumab dose B.
  Interventions: Drug: Risankizumab Dose B

INTERVENTIONS:
Drug: Risankizumab Dose A — Prefilled Syringe
  Arms: Risankizumab Dose A
Drug: Risankizumab Dose B — Prefilled Syringe
  Arms: Risankizumab Dose B

SUMMARY:
This study will assess how safe risankizumab is and how risankizumab moves through the body of adult healthy participants. Adverse Events will be assessed.

Risankizumab is an investigational drug being developed for the treatment of Crohn's Disease. Participants are randomly assigned to one of the 2 treatment groups. Approximately 198 adult healthy volunteers will be enrolled in at least 4 sites across the world.

All participants will receive risankizumab as subcutaneous injections in one of the 2 different formulations.

There may be higher burden for participants in this trial. Participants will be confined for 10 days and followed up for 140 days. Adverse Events and blood tests will be collected.

ELIGIBILITY:
Inclusion Criteria:

- Body weight greater than 40 kg and less than 100 kg at screening and upon initial confinement.

Exclusion Criteria:

* Previous exposure to any anti-interleukin-12/23 or anti-interleukin-23 treatment.
* Intention to perform strenuous exercise to which the participant is unaccustomed within one week prior to administration of study drug or during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Approximately up to 113 days
  Maximum Observed Plasma Concentration (Cmax)
Time to Maximum Observed Plasma Concentration (Tmax) | Approximately up to 113 days
  Time to Maximum Observed Plasma Concentration (Tmax)
Apparent Terminal Phase Elimination Rate Constant (β) | Approximately up to 113 days
  Apparent Terminal Phase Elimination Rate Constant (β)
The Terminal Phase Elimination Half-Life (t1/2) | Approximately up to 113 days
  The Terminal Phase Elimination Half-Life (t1/2)
The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt) | Approximately up to 113 days
  The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt)
The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC∞) | Approximately up to 113 days
  The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC∞)
Number of Participants with Adverse Events | Approximately up to 140 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (5):
- United States (5):
  - Anaheim Clinical Trials LLC /ID# 250098, Anaheim, California
  - Clinical Pharmacology of Miami /ID# 250099, Miami, Florida
  - Acpru /Id# 249681, Grayslake, Illinois
  - Bio-Kinetic Clinical Applications, LLC /ID# 250181, Springfield, Missouri
  - PPD Clinical Research Unit - Austin /ID# 250672, Austin, Texas

IPD SHARING:
Plan to Share IPD: No